CLINICAL TRIAL: NCT04896710
Title: Rapid Testing for Self-Administration Among an Asymptomatic Sample
Brief Title: COVID-19 Rapid Testing for Self-Administration Among an Asymptomatic Sample
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of British Columbia (Other)
Collaborators: Health Canada (Other Government); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Sabrina Wong, PhD, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 331297
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Asymptomatic Shedding Viral
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self administration (Experimental): The participant will self administer the SD Biosensor. Their rapid antigen test result will be compared to health care professional administered SD Biosensor
  Interventions: Device: SD Biosensor

INTERVENTIONS:
Device: SD Biosensor — Nasal swab SD biosensor to be self administered

SUMMARY:
Point-of-care testing can provide an additional layer of protection to reduce transmission of COVID-19 safely and effectively in the population, and if such tests can be self-administered, barriers to access may be reduced. The investigators will conduct a study among those self-identifying as asymptomatic for COVID-19 to evaluate the reliability and feasibility of self-administration of a point-of-care nasal swab test, determine the sensitivity and specificity of the point-of-care nasal swab test relative to reverse transciptase polymerase chain reaction (RT-PCR) testing, and gather quantitative and qualitative data on the acceptability and self efficacy of self-administration.

DETAILED DESCRIPTION:
In Canada, the age distribution of COVID-19 has demonstrated that young adults are susceptible to infection. As of mid-December, about 19% of cases have occurred in the 20-29 year age group, and about 3% of those hospitalized were 20-29 years of age. In BC, in week 50, the incidence was highest in adults 20-29 years (127 cases per 100,000 population), which is four times higher than what was observed in week 38 (30 cases per 100,000 population). These statistics highlight the need to disrupt transmission in this group.

Congregate living settings have been established as high-risk environments for community transmission of SARS-CoV-2. Moreover, there is a need to ensure the workforce feels safe in returning back to work across post-secondary institutions. While the COVID-19 vaccine rollout has commenced in BC, according to experts in the field, the pandemic is likely to persist for some time. For people living in congregate housing and for post-secondary institutions to open safely, COVID-19 mitigation strategies are as important as ever. There is no current public health strategy used for systematic COVID-19 screening for those living in congregate housing. Individuals are expected to monitor themselves daily for symptoms and use "multiple layers of protection" which include physical distancing, mask wearing and hand washing.

However, this strategy is not very effective because these measures are relatively insensitive and thus unlikely to identify all individuals with SARS-CoV2, especially those who are minimally symptomatic or believe they are asymptomatic. Indeed, public health experts have poignantly stated that transmission of the virus through asymptomatic individuals is the "Achilles' Heel of Current Strategies to Control COVID-19" (1). This is because, unlike SARS-CoV-1, the cause of the original SARS epidemic in 2003, SARS-CoV-2 sheds at high concentrations from the nasal cavity even in asymptomatic individuals, who may harbour the virus but have yet to demonstrate any symptoms during the prodromal phase of the disease (2). Even with masking and social distancing, such individuals could be at a high risk of spreading the virus in congregate housing and in enclosed spaces (e.g. classrooms). One approach to reducing the risk of SARS-CoV-2 transmission amongst those living in congregate housing and working in enclosed spaces with large numbers of people (e.g. classrooms) is to "screen" for those who are likely to harbour the virus (even though they may have no or minimal symptoms). However, the current diagnostic approach, which uses real-time reverse transcriptase polymerase chain reaction (RT-PCR) to detect the presence of viral RNA from nasopharyngeal swabs, cannot be easily deployed for this purpose.

The RT-PCR test is expensive (>$100/test), time-consuming (with turnaround times of 1-2 days) and requires trained healthcare personnel to administer the test. A potential solution to this conundrum is to use a "point-of-care" test, which can be deployed at either work or a congregate housing site and whose results will be available within one hour of testing. However, for these assays or platforms to be viable, they will need to be used as "screening" rather than "diagnostic" tests (see below for more detailed discussion on this topic), and be relatively simple to use (so ideally they can be self-administered) and inexpensive.

What is the difference between diagnostic and screening tests?

Diagnostic testing for SARS-CoV-2 is intended to identify occurrence at the individual level and is performed when there is a reason to suspect that an individual may be infected, such as having symptoms or suspected recent exposure, or to determine resolution of infection. Examples of diagnostic testing include testing symptomatic individuals who present to their healthcare provider, testing individuals through contact tracing efforts, testing individuals who indicate that they were exposed to someone with a confirmed or suspected case of COVID-19, and testing individuals present at an event where an attendee was later confirmed to have COVID-19. The U.S. Food and Drug Administration's (FDA) FAQs on Testing for SARS-CoV-2 also address diagnostic testing for SARSCoV-2.

Screening tests for SARS-CoV-2, on the other hand, are intended to identify occurrence at the individual level even if there is no reason to suspect infection-e.g., there is no known exposure. This includes, but is not limited to, screening of asymptomatic individuals without known exposure with the intent of making decisions based on the test results. Screening tests are intended to identify infected individuals without, or prior to development of, symptoms who may be contagious so that measures can be taken to prevent further transmission. Examples of screening include testing plans developed by a workplace to test its employees, and testing plans developed by a school to test its students, faculty, and staff. In both examples, the intent is to use the screening testing results to determine who may continue to participate in activities and the protective measures that must be taken, including self-isolation. FDA's FAQs on Testing for SARSCoV- 2 also address screening testing for SARS-CoV-2.

In summary, a screening COVID-19 test is one that is specific for SARS-CoV-2 but has a lower sensitivity (i.e., ability to detect the virus) than that of a diagnostic test (the gold standard). Thus, even those who have a negative screening test should be considered potentially infectious and must adhere to social distancing, masking rules and all other public health orders/guidelines. Those who are tested positive on the screening test must be assumed to have COVID-19 until proven otherwise by a confirmatory RT-PCR test. This approach of using "point-of-care" screening tests was recently advocated by The New England Journal of Medicine (3).

The investigators have conducted a feasibility pilot from February 9-April 23, 2021 at Orchard Commons, University of British Columbia. The investigators tested BD Veritor nasal swab rapid antigen test since it was already approved by Health Canada and supported by the Vancouver Coastal Health Medical Health Officer. The investigators examined the feasibility of participants to self-collect nasal swabs and considered the ability to complete the rapid antigen test. The BD Veritor system entails much accuracy of putting the mucosal cells into the small dropper. This system also has an analytic reader. The investigators believe this system will be useful when it can be administered by a trained person because of the dropper and the need for an analytic reader. Based on a small survey (n=184), the team concluded that following:

Nasal swabs are acceptable (99% of participants rated nasal swabbing as acceptable/very acceptable).

Rapid antigen tests need to take no longer than 15 minutes. In order to move to self administration, the team believes there should be no analytic reader and that the participant should be able to tell with a visual examination if the rapid antigen test was positive (much like a pregnancy test). The Roche SD biosensor test was chosen for this study since it is a low complexity test that can likely be used by many of the general public.

Primary Goal: The primary goal of this study is to determine and test the feasibility, reliability, and sensitivity/specificity of COVID-19 self-administered screening amongst those who are asymptomatic and living and/or working at UBC. The investigators will evaluate whether rapid antigen testing can identify virus transmission chains early through the identification of pre-symptomatic and asymptomatic cases, and direct students and staff with positive test results to follow appropriate public health precautions - all of which are proven to minimize viral spread.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 16 years and over
* Living or working at University of British Columbia
* Self identified as asymptomatic for COVID-19
* Participants able to give written informed consent

Exclusion Criteria:

* Anyone who is self identified as having COVID-19 symptoms
* Those diagnosed with COVID-19 in last 30 days

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 569 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Concordance | 2 months
  Concordance (calculated using Cohen's Kappa) between self administered and health care professional administered SD Biosensor rapid antigen test results.
Ability of rapid antigen test to detect COVID-19 positive | 3 months
  >80% sensitivity and >95% specificity for SD Biosensor rapid antigen test among asymptomatic population

SECONDARY OUTCOMES:
Acceptability of self administration | 3 months
  Self reported acceptability of self administration will be collected from participants by questionnaire; acceptability will be defined by 4 response categories: very acceptable, acceptable, somewhat acceptable, not at all acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina T Wong, RN, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Orchard Commons, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
A de-identified and anonymized dataset can be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: August 31, 2022
Access Criteria: send email to: jonathan.beaumier@ubc.ca

REFERENCES:
- [Background] Gandhi M, Yokoe DS, Havlir DV. Asymptomatic Transmission, the Achilles' Heel of Current Strategies to Control Covid-19. N Engl J Med. 2020 May 28;382(22):2158-2160. doi: 10.1056/NEJMe2009758. Epub 2020 Apr 24. No abstract available. PMID 32329972
- [Background] Arons MM, Hatfield KM, Reddy SC, Kimball A, James A, Jacobs JR, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Dyal JW, Harney J, Chisty Z, Bell JM, Methner M, Paul P, Carlson CM, McLaughlin HP, Thornburg N, Tong S, Tamin A, Tao Y, Uehara A, Harcourt J, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Montgomery P, Stone ND, Clark TA, Honein MA, Duchin JS, Jernigan JA; Public Health-Seattle and King County and CDC COVID-19 Investigation Team. Presymptomatic SARS-CoV-2 Infections and Transmission in a Skilled Nursing Facility. N Engl J Med. 2020 May 28;382(22):2081-2090. doi: 10.1056/NEJMoa2008457. Epub 2020 Apr 24. PMID 32329971
- [Background] Mina MJ, Parker R, Larremore DB. Rethinking Covid-19 Test Sensitivity - A Strategy for Containment. N Engl J Med. 2020 Nov 26;383(22):e120. doi: 10.1056/NEJMp2025631. Epub 2020 Sep 30. No abstract available. PMID 32997903